CLINICAL TRIAL: NCT05745168
Title: Pilot Implementation of HIV Self-testing Delivery in Private Pharmacies Combined to a Respondent Driven Sampling Method to Improve HIV Testing for MSM and TGW in Phnom Penh - ANRS 0100s
Status: Not yet recruiting | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Saglik Bilimleri Universitesi (Other); Sciences économiques et sociales de la santé et traitement de l'information médicale Marseille France (Unknown); National Center For HIV/AIDS, DERMATOLOGY AND STD Phnom Penh, Cambodia (Unknown); Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS0100s
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: HIV Infections
Keywords: Self-testing; Private pharmacy; RDS; MSM; Transgender women
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSM-TGW
  Interventions: Diagnostic Test: OraQuick

INTERVENTIONS:
Diagnostic Test: OraQuick — The intervention is based on respondent-driven sampling approach. Each selected seed from hotspots and on social networks is provided with two types of coupons for HIVST kit at partner pharmacy: electronic coupons (e-coupons) consisting of a pictured unique anonymous QR code and identifier and the address of pharmacies; paper coupons consisting of similar information to e-coupon. The seeds will then distribute coupons to their networks physically, via social media, and smart phone applications. Each recruited participant will bring the coupon to be scanned at the pharmacies to receive a free access HIVST kit. There, trained community worker will do the study visit including information/consent, e-CRF filling and providing link to send the test results. These recruited individuals will be considered as wave 1 and will each receive 10 additional coupons to recruit new members in the networks. The next round of individuals recruited and enrolled will be considered as wave 2, and so on.

SUMMARY:
The study aims to evaluate the feasibility of HIV self-testing (HIVST) delivery by a private pharmacy network among men who have sex with men (MSM) and transgender women (TGW) recruited through a classic and digital Respondent Driven Sampling method to improve HIV testing in Phnom Penh, Cambodia.

An interventional pilot study using a mixed qualitative and quantitative approach will be carried out in order to evaluate the feasibility, acceptability and appropriateness of the strategy and to identify barriers and facilitators.

DETAILED DESCRIPTION:
INTRODUCTION AND OBJECTIVES

The last Cambodian 2019 IBBS report highlighted the fact that half of men who have sex with men (MSM) and one third of transgender women (TGW) were never tested for HIV or since more than 12 months. Receiving HIV education and materials in the past 6 months and perception of higher HIV risk compared to the general population were the common factors associated with the increasing HIV testing uptake. In this report, the majority of MSM and TGW were tested at Community-based organizations (CBO) facilities and by CBO outreach workers while private facilities are poorly used for HIV testing (5% for MSM and 2% for TGW). Private pharmacies could be able to deliver HIV selftesting (HIVST) kits giving the advantage of confidentiality, anonymity and time-saving, in particular for those reluctant to visit CBOs by lack of secrecy regarding their sexual orientation.The recruitment of participants by RDS could give the opportunity to reach MSM and TGW outside the network of CBOs.

The principal objective is to evaluate the feasibility of HIV self-testing (HIVST) delivery by a private pharmacy network among men who have sex with men (MSM) and transgender women (TGW) recruited through a classic and digital Respondent Driven Sampling method to improve HIV testing in Phnom Penh, Cambodia

Our secondary objectives are:

* Evaluate the acceptability and appropriateness of the strategy
* Identify barriers and facilitators
* Estimate the linkage to confirmatory testing for those with a reactive test and linkage to HIV care and ART for those with a positive confirmatory HIV test
* Estimate linkage to pre-exposure prophylaxis (PrEP) services for negative participants
* Estimate the characteristics of participants and compare to those reported in Integrated Biological and Behavioral Survey (IBBS 2019) for MSM and TGW in Cambodia
* Evaluate the adherence of participants to a 6-monthly repeated HIV testing

METHODOLOGY

Study design An interventional pilot study using a mixed qualitative and quantitative approach will be carried out in order to evaluate the feasibility, acceptability and appropriateness of the strategy and to identify barriers and facilitators.

The participant recruitment method will be designed as a Respondent Driven Sampling (RDS) by recruiting initial seeds both at hotspots and on social networks.

After 6 months, a qualitative assessment by focus groups discussion (FGD) will be conducted among MSM, TGW and pharmacists to evaluate feasibility, acceptability and appropriateness of the intervention and to identify barriers and facilitators.

Each participant will be followed during 18 months and encouraged to perform a 6-monthly HIV testing during this period.

Study overview

The intervention will be designed as a RDS by recruiting initial seeds both at hotspots and on social networks. 15 initial seeds will be recruited. Seeds will come to the study site for checking inclusion criteria and receiving information on self-testing, benefits of their participation and recruiting other participants in their networks along with the important details about the study. Once consent to the study, the seed is provided with two types of coupons for HIVST kit at partner pharmacy: 5 electronic coupons (e-coupons) consisting of a pictured unique anonymous QR code and identifier and address of partner pharmacies; 5 paper coupons consisting of a printed unique anonymous QR code, identifier and address of partner pharmacies. The seeds will then distribute electronic and paper coupons to their networks physically and via social media, messaging and calling applications such as Twitter, Whatapp and Telegram (e-coupons).

Each recruited participant will bring the coupon to be scanned at partner pharmacies to receive direct and free access to one HIVST kit. Partner pharmacies with a proper dedicated room/space securing privacy and secrecy in Phnom Penh are the study sites. There, trained community worker/research team who get notified by partner at each visit of participant will do the study visit including information/consent, e-CRF filling and give a link of an external website to send the HIV test results and receive information or advices.

These recruited individuals will be considered as wave 1 of recruitment and will each receive 10 additional coupons to recruit the members of their networks. The next round of individuals recruited and enrolled will be considered as wave 2, and so on. The number of 10 coupons was selected to avoid a bias risk related to participation incentives.

To facilitate the return of HIVST kit results, participant will upload the picture of results labeled with their identifier directly using the link of the external website that they received from community worker/research team during their visits at pharmacy. In case of any question, they could reach community worker/research team by hotline number. According to the results, the participants will be proposed with a support for linkage to confirmatory test or to PrEP services. Each non-reactive participant will be provided another new coupon (paper or electronic format upon their preference) with a reminder to perform a 6-monthly HIV testing during 18 months. They will not be granted any token or incentives if they fail to return the result of HIVST kit taken at pharmacies.

After 6 months, a qualitative assessment will be conducted to evaluate feasibility, acceptability and appropriateness of the intervention and to identify barriers and facilitators.

Several ART sites/HIV clinics particularly in charge of key populations will be specifically selected as participating centers in order to collect information on linkage to care or prevention services for positive and negative participants, respectively.

Statistical methods

To evaluate the feasibility of the intervention to improve HIV testing among MSM and TGW in Phnom Penh, a pragmatic approach with the objective to recruit the maximum of MSM and TGW was carried out. According to the IBBS 2019, the estimated number of MSM in Phnom Penh is 6300 and the estimated number of TGW is 1400.

With 1500 participants (1000 MSM and 500 TGW), the proportion of an HIV self-test uptake was estimated to be 70% to within a 95% confidence interval of +/- 2 - 2.5% (width of the confidence interval (in %) = 1.96 x √( p x (1-p) / n)). Intervention

RDS intervention

The seeds will be recruited at hotspots, online applications and social media networks. Hotspots include steam sauna and spa and gay bars and clubs. Online applications and social media include Facebook groups, twitter, telegram, whatapps and other date applications such as Grindr, Planet Romeo, Hornet, Blued.

Prior to seed recruitment, a consultative meeting will be conducted among pimps (a person who controls sex workers, especially by finding customers for them, and takes some of the money that they earn), procurers (a person who finds sex workers for people who want to have sex with them), high class MSM & TGW, network organizers, social media group organizers in order to optimize the selection criteria of the seeds.

Selection criteria obtained from the meeting with pimps, procurers, high class MSM, network organizers, twitter groups organizer is applied to select the initial seeds that are very likely to lead us to reach a large diversity of MSM&TGW population.

A number of 15 seeds will be selected firstly to ensure the representation of gender, age group, sexual behaviors, and participation in sex work. If necessary, new seeds could be recruited later. Seeds will come to the study site for checking inclusion criteria and receiving information on self-testing, benefits of their participation and recruiting other participants in their networks along with the important details about the study. Once consent to the study, the seed is provided with two types of coupons for HIVST kit at partner pharmacy: 1- 5 electronic coupons (e-coupons) consisting of a pictured unique anonymous QR code and identifier and address of partner pharmacies 2- 5 paper coupons consisting of a printed unique anonymous QR code, identifier and address of partner pharmacies. The seeds will provide paper- and e-coupons to their networks physically and via social media, messaging and calling applications such as Twitter, Whatapp and Telegram (e-coupons). For online application and social media, a peer could be reached by chat or call.

When the participant arrives in a partner pharmacy, the coupon (unique QR code with identifier) will be scanned by the pharmacist prior to the free delivery of HIV self-test. Community workers (CWs) will be then alerted by the pharmacist for study visits to participant directly at the dedicated space at the pharmacy. During the visit with CW, participant will receive the information about the study, check for eligibility criteria, ask to be recontacted by phone and participation in FGD, fill in the detailed e-CRF, receive the information on HIV self-testing instructions, list of partner pharmacies, helpline phone number, location of the 2 partners ART sites, location of the HIV clinics with prevention services and PrEP delivery availability, be provided one free HIV self-testing kit delivered Incentives will be provided in two steps for participants to encourage them to return the results of HIVST and recruit their peers. In step one, each participant will receive 2 USD for returning the HIVST result successfully to the provided link. In step two, an amount of 1 USD will be provided for each recruited peer. This amount was decided as a balance between feasibility (encouragement) and sustainability of the strategy (not too high for possible scaling-up).

In case of any issue for tablet use or HIVST kit use, helpline phone number will be available. One dedicated community worker funded by the study will be in charge to manage helpline service.

Intervention after delivering HIV test result

In case of reactive HIV test, the participant could join immediately one research team by hotline or messages on the website that will provide support and orientation. After 1 week, contact with the participant will be done by phone by the research team (if the participant gave consent) to confirm the linkage to one of the partner ART sites. The linkage between participants and HIV clinics will be done by the initial QR code.

If the linkage to confirmatory testing and/or care is not confirmed, a community worker provides additional assistance to the participants.

In case of non-reactive test, the participant could download in the external website one electronic coupon (QR code) to repeat the HIV test 6 month later. Participants will be informed on the external website about the possibilities to join the pilot PrEP program in Chhouk Sar clinic in Phnom Penh.

Qualitative assessment

After 6 months, a qualitative assessment will be conducted to evaluate acceptability and appropriateness of the intervention. Qualitative assessment will be done by focus groups. Focus groups will be conducted in 3 specific populations: MSM, TGW and pharmacists. For each population of MSM and TGW, a qualitative sample will be selected in order to capture different profiles according to sex behaviors and demographic and socioeconomic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* To be aged from 18 years old (legal age in Cambodia)
* For MSM, to have at least one oral or anal intercourse with another man in the past 12 months
* For TGW, to be biologically a male at birth and self-identified as a woman or third gender and have at least one oral, anal or vaginal intercourse with another man in the past 12 months

Exclusion Criteria

* Known HIV positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For MSM, to have at least one oral or anal intercourse with another man in the past 12 months; For TGW, to be biologically a male at birth and self-identified as a woman or third gender and have at least one oral, anal or vaginal intercourse with another man in the past 12 months
Study Population: The survey population consists of MSM and TGW aged from 18 years old who are living in Phnom Penh at the study period regardless of their nationalities or migration history (moving from other provinces)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability proportion of HIV self-test by MSM/TGW provided by private pharmacy | February 2023 to April 2025
  Number of HIV self-tests delivered / total number of coupons distributed

SECONDARY OUTCOMES:
Acceptability and appropriateness provision of HIV self-test to MSM/TGW via private pharmacy | February 2023 to April 2025
  Group discussion using topic guides focusing on the comfortability, usefulness, suitability, confidentiality, credibility, advantages and barriers of provision of HIV self-test to MSM/TGW via private pharmacy among participants and private pharmacies

CONTACTS AND LOCATIONS:
Overall Officials: Vonthanak Saphonn, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Mohamed Ben-Mechlia, PhD, Study Director — ANRS, Emerging Infectious Diseases; Bruno Spire, PhD, Principal Investigator — SESSTIMS
Locations (1):
- University of Health Sciences, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dary C, Segeral O, Larmarange J, Mosnier E, Ben Mechlia M, Ouk V, Spire B, Saphonn V. Pilot Implementation of HIV Self-Testing Delivery in Private Pharmacies Combined With a Respondent-Driven Sampling Method to Improve HIV Testing for Men Who Have Sex With Men and Transgender Women in Phnom Penh (ANRS 0100s): Protocol for a Prospective Mixed Method Feasibility Study. JMIR Res Protoc. 2025 Jun 27;14:e65351. doi: 10.2196/65351. PMID 40577719

DOCUMENTS (1):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT05745168/Prot_001.pdf